CLINICAL TRIAL: NCT03407482
Title: A Phase II, Open-Label Extension Study of Patients Previously Enrolled in Study GA30044 to Evaluate the Long-Term Safety and Efficacy of GDC-0853 in Patients With Moderate to Severe Active Systemic Lupus Erythematosus
Brief Title: An Extension Study of GDC-0853 in Participants With Moderate to Severe Active Systemic Lupus Erythematosus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was ended early due to the lack of efficacy seen in the parent study GA30044.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA30066; 2017-001764-37 (EudraCT Number)
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — fenebrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GDC-0853 (200mg) BID (Experimental): Participants previously enrolled in the parent GA30044 Study, now received GDC-0853 (200mg) orally twice daily (BID).
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — Participants received GDC-0853 at a dose of 200mg, as per the dosing schedule described above.

SUMMARY:
This Phase II, multicenter, open-label extension (OLE) study will evaluate the long-term safety and efficacy of GDC-0853 in participants with systemic lupus erythematosus (SLE) who have completed Study GA30044 (NCT02908100) up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to comply with the study protocol, in the investigator's judgment
* Completion of Study GA30044 up to 48 weeks
* Acceptable safety and tolerability during Study GA30044 as determined by the investigator

Exclusion Criteria:

* Met protocol-defined treatment-stopping criteria during Study GA30044
* An adverse event in Study GA30044 that required permanent discontinuation of study drug
* In the opinion of the investigator, any new, significant, uncontrolled comorbidity or new clinical manifestation (related to SLE or not) that requires medications not allowed in this protocol; or could put the participant at undue risk from a safety perspective
* Any uncontrolled or clinically significant laboratory abnormality that would affect safety, interpretation of study data, or the participant's participation in the study in the opinion of the investigator in consultation with the Medical Monitor

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- United States (10):
  - Valerius Medical Group, Los Alamitos, California
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - Tekton Research Inc, Austin, Texas
  - Accurate Clinical Research, Houston, Texas
  - Arthritis Clinic Of Central Texas, San Marcos, Texas
- Argentina (4):
  - APRILLUS, Buenos Aires
  - Hospital Italiano de La Plata, La Plata
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Médico Privado de Reumatología, San Miguel de Tucumán
- Brazil (9):
  - CIP - Centro Internacional de Pesquisa, Goiânia, Goiás
  - Centro Mineiro de Pesquisa - CMIP, Juiz de Fora, Minas Gerais
  - Edumed - Educação e Saúde SA, Curitiba, Paraná
  - Centro de Pesquisas em Diabetes - CPD, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC*X*, Santo André, São Paulo
  - Centro de Pesquisas Clinicas; CPCLIN, São Paulo, São Paulo
  - Hospital Abreu Sodré - AACD, São Paulo, São Paulo
- Bulgaria (6):
  - MHAT Plovdiv, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - Medical Center Excelsior OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Chile (4):
  - CTR Estudios SPA, Providencia
  - Dermacross, Santiago
  - Centro de Estudios Reumatologi, Santiago
  - Biomedica, Santiago
- Colombia (5):
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Barranquilla
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Medicity S.A.S., Bucaramanga
  - Servimed S.A.S., Bucaramanga
  - Hospital Pablo Tobon Uribe, Medellín
- Mexico (5):
  - Centro de Investigacion Alberto Bazzoni S.A. de C.V., Torreón, Coahuila
  - Unidad de Atencion Medica e Investigacion en Salud S.C., Mérida, Yucatán
  - Hospital Angeles Lindavista, México
  - Hospital Universitario de Saltillo, Saltillo
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosi S.l.p.
- Konkuk University Medical Center, Seoul, South Korea
- Spain (5):
  - Fundación Profesor Novoa Santos, A Coruña, LA Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico Universitario Valladolid, Valladolid
  - Hospital Universitario Rio Hortega, Valladolid
- Taiwan (2):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Guy's Hospital; Louise Coote Lupus Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 50 centers in 11 countries.
Pre-assignment Details: 160 participants were enrolled into this OLE study and were included in the ITT and Safety populations.
Period: Overall Study
Arm/Group | GDC-0853 (200mg) BID
Started | 160
Completed | 29
Not Completed | 131
Not completed — Adverse Event | 12
Not completed — Disease Relapse | 1
Not completed — Lost to Follow-up | 1
Not completed — Non-Compliance With Study Drug | 1
Not completed — Pregnancy | 2
Not completed — Protocol Violation | 1
Not completed — Study Terminated By Sponsor | 106
Not completed — Withdrawal by Subject | 6
Not completed — Data Entry Error | 1

BASELINE CHARACTERISTICS:
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 5
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 117
    Not Hispanic or Latino | 42
    Not Stated | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    American Indian or Alaska native | 24
    Asian | 5
    Black or African American | 22
    Multiple | 5
    White | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: Baseline up until 8 weeks after the last dose of study drug (up to 56 weeks)
Population: The Safety-evaluable population was defined as all participants who received at least one dose of the study drug during this OLE study.
Measure: Number; unit: Percentage of Participants
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 160
Percentage of Participants | 64.4

2. Secondary Outcome: Systemic Lupus Erythematosus Responder-4 Index (SRI-4) up to Week 48
Description: The Systemic Lupus Erythematosus Responder Index (SRI)-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Baseline up to Week 48
Population: Please note that for this Outcome Measure, no data was collected at all due to no participants being evaluated at all, as a result of early termination of this study due to fenebrutinib not demonstrating improved efficacy compared to placebo across secondary or exploratory endpoints in the parent study (Study GA30044).
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 0

3. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time t (AUC0-t,ss) of GDC-0853 at Steady State
Description: Population PK model estimated AUC of GDC-0853 From Time 0 to Time t (AUC0-t) at steady-state. AUC was measured in Nanograms (ng) per millilitre(mL)*hour (hr).
Time Frame: Pre-dose (0 hour [hr]) at Weeks 0, 24, 48, at unscheduled or flare or early termination visit (up to Week 56)
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (AUC0-t,ss) parameter could not be generated via the Population PK model.
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 0

4. Secondary Outcome: Minimum Plasma Concentration of GDC-0853 at Steady State (Ctrough,ss)
Description: Population PK model estimated minimal plasma concentration (Ctrough) of GDC-0853 at steady-state (ss).
Time Frame: Pre-dose (0 hr) at Weeks 0, 24, 48, at unscheduled or flare or early termination visit (up to Week 56)
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (Ctrough,ss) parameter could not be generated via the Population PK model.
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 0

5. Secondary Outcome: Plasma Decay Half-Life of GDC-0853 at Steady State (t1/2,ss)
Description: Population PK model estimated plasma decay half life of GDC-0853 at steady-state.
Time Frame: Pre-dose (0 hr) at Weeks 0, 24, 48, at unscheduled or flare or early termination visit (up to Week 56)
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (t1/2,ss) parameter could not be generated via the Population PK model.
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 0

6. Secondary Outcome: Apparent Oral Clearance of GDC-0853 at Steady State (CL/F,ss)
Description: Population PK model estimated apparent oral clearance of GDC-0853 at steady-state.
Time Frame: Pre-dose (0 hr) at Weeks 0, 24, 48, at unscheduled or flare or early termination visit (up to Week 56)
Population: Please note that for this Outcome Measure, incomplete PK data was collected as a result of early termination of the study which meant that data for the (CL/F,ss) parameter could not be generated via the Population PK model.
Arm/Group | GDC-0853 (200mg) BID
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up until 8 weeks after the last dose of study drug (up to 56 weeks)
Arm/Group | GDC-0853 (200mg) BID
All-Cause Mortality (participants affected / at risk) | 0/160
Serious Adverse Events (participants affected / at risk) | 4/160
Other Adverse Events (participants affected / at risk) | 31/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0853 (200mg) BID (N=160)
CELLULITIS (Infections and infestations) | 1 (1)
INFECTIVE TENOSYNOVITIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0853 (200mg) BID (N=160)
NAUSEA (Gastrointestinal disorders) | 9 (9)
NASOPHARYNGITIS (Infections and infestations) | 13 (14)
URINARY TRACT INFECTION (Infections and infestations) | 15 (15)

LIMITATIONS AND CAVEATS:
The study was ended early due to the lack of efficacy seen in the parent study GA30044.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03407482/Prot_SAP_000.pdf